CLINICAL TRIAL: NCT01583127
Title: Examining Variation in the Impact of School-Wide Positive Behavioral Interventions and Supports (PBIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H.33.02.03.07.A; R01MH067948 (NIH)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Problem Behavior
Keywords: Problem Behavior
MeSH Terms: conditions — Problem Behavior | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- School-Wide (SW)-PBIS intervention (Experimental): SW-PBIS intervention
  Interventions: Behavioral: Positive Behavioral Interventions & Supports
- Control (No Intervention): Practice as usual

INTERVENTIONS:
Behavioral: Positive Behavioral Interventions & Supports — Implementation of the School-Wide Positive Behavioral Interventions and Supports model across 4 school years.
  Other Names: Positive Behavior Supports
  Arms: School-Wide (SW)-PBIS intervention

SUMMARY:
To conduct a randomized controlled trial of School-Wide Positive Behavioral Interventions and Supports, which is a school-based prevention program aimed at reducing behavior problems in children.

DETAILED DESCRIPTION:
To conduct a group randomized controlled trial of School-Wide Positive Behavioral Interventions and Supports. PBIS is a popular school-based prevention program aimed at reducing behavior problems in children. Staff are trained to implement behavioral focused prevention programs to address issues related to student conduct and discipline problems.

ELIGIBILITY:
Inclusion Criteria:

* Public Elementary Schools
* All children attending the schools and staff employed were eligible for inclusion

Exclusion Criteria:

• None

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32986 (Actual)
Dates: Start 2002-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Teacher ratings | 5 time points over 4 years
  teacher ratings of students prosocial behavior, emotion regulation, conduct problems, and aggressive behavior

SECONDARY OUTCOMES:
student discipline data | 5 time points over 5 years
  suspensions, office discipline referrals
school climate | 5 time points over 5 years
  teacher and student reports of school climate

CONTACTS AND LOCATIONS:
Overall Officials: Catherine P Bradshaw, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Result] Bradshaw CP, Pas ET, Bloom J, Barrett S, Hershfeldt P, Alexander A, McKenna M, Chafin AE, Leaf PJ. A state-wide partnership to promote safe and supportive schools: the PBIS Maryland Initiative. Adm Policy Ment Health. 2012 Jul;39(4):225-37. doi: 10.1007/s10488-011-0384-6. PMID 22246614
- [Result] Bradshaw CP, Koth CW, Thornton LA, Leaf PJ. Altering school climate through school-wide Positive Behavioral Interventions and Supports: findings from a group-randomized effectiveness trial. Prev Sci. 2009 Jun;10(2):100-15. doi: 10.1007/s11121-008-0114-9. PMID 19011963
- [Result] Bradshaw, C. P., Mitchell, M. M., & Leaf, P. J. (2010). Examining the effects of School-Wide Positive Behavioral Interventions and Supports on student outcomes: Results from a randomized controlled effectiveness trial in elementary schools. Journal of Positive Behavior Interventions, 12, 133-148.
- [Result] Bradshaw, C.P., Koth, C.W., Bevans, K.B., Ialongo, N., & Leaf, P.J. (2008). The impact of school-wide Positive Behavioral Interventions and Supports (PBIS) on the organizational health of elementary schools. School Psychology Quarterly, 23(4), 462-473.
- [Result] Waasdorp TE, Bradshaw CP, Leaf PJ. The impact of schoolwide positive behavioral interventions and supports on bullying and peer rejection: a randomized controlled effectiveness trial. Arch Pediatr Adolesc Med. 2012 Feb;166(2):149-56. doi: 10.1001/archpediatrics.2011.755. PMID 22312173
- [Derived] Stuart EA, Bradshaw CP, Leaf PJ. Assessing the generalizability of randomized trial results to target populations. Prev Sci. 2015 Apr;16(3):475-85. doi: 10.1007/s11121-014-0513-z. PMID 25307417
- [Derived] Bradshaw CP, Waasdorp TE, Leaf PJ. Effects of school-wide positive behavioral interventions and supports on child behavior problems. Pediatrics. 2012 Nov;130(5):e1136-45. doi: 10.1542/peds.2012-0243. Epub 2012 Oct 15. PMID 23071207